CLINICAL TRIAL: NCT04915313
Title: The Antihypertensive Effect of Remote Ischemic Conditioning: A Multicenter, Randomized, Double-blind, Sham-controlled Trial.
Brief Title: The Antihypertensive Effect of Remote Ischemic Conditioning (RIC-HTN).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Peking University Care Health Management Center (Unknown); The 306 Hospital of People's Liberation Army (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIC-HTN
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Hypertension,Essential; Prehypertension
Keywords: Remote ischemic conditioning; Essential hypertension; Prehypertension; Blood pressure
MeSH Terms: conditions — Essential Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in the intervention group will recieve remote ischemic conditioning (RIC) treatment twice a day for 4 weeks.
  Interventions: Device: Remote ischemic conditioning (RIC)
- Sham control group (Sham Comparator): Subject in the sham control group will recieve sham remote ischemic conditioning (Sham-RIC) treatment twice a day for 4 weeks..
  Interventions: Device: Sham remote ischemic conditioning (Sham-RIC)

INTERVENTIONS:
Device: Remote ischemic conditioning (RIC) — RIC is a non-invasive therapy which is performed by automated pneumatic cuffs placed on bilateral arms. The RIC protocol include five cycles of 5-min inflation to 200mmHg and 5-min deflation.
  Arms: Intervention group
Device: Sham remote ischemic conditioning (Sham-RIC) — The Sham-RIC protocol include five cycles of 5-min inflation to 60 mmHg and 5-min deflation by placing automated pneumatic cuffs on bilateral arms.
  Arms: Sham control group

SUMMARY:
This study intends to further reveal the antihypertensive effect of LRIC and explore its potential mechanisms.

DETAILED DESCRIPTION:
Stroke is the second-leading cause of death in the world and the leading cause of death in China. The estimated lifetime risk of stroke for those aged 25 years old and above is 24.9% worldwide and 39.3% in China. Hypertension is one of the main independent risk factors for stroke. Studies have shown that the risk of stroke increase at blood pressure (BP) above 115/75mmHg, each increase of 20mmHg in systolic blood pressure (SBP) or 10 mmHg in diastolic blood pressure (DBP) will double the risk of stroke. For those hypertensive patients without complications, each reduction of 10mmHg in SBP reduces approximately 17% risk of stroke, and each reduction of 5mmHg in DBP reduces 20%. Therefore, enhancing the primary prevention of stroke in hypertensive patients without vascular complications is important to reduce the burden of stroke in the future. However, these patients do not pay enough attention to their elevated BP and have poor compliance with antihypertensive drugs. Therefore, it is necessary to explore an economical, convenient and effective non-pharmacological therapy to control BP in order to reduce the risk of stroke.

Limb remote ischemic conditioning (LRIC) triggers endogenous protective effect through transient and repeated ischemia in the limb to protect remote tissues and organs. The mechanisms of LRIC involve the regulation of autonomic nervous system, release of humoral factors, improvement of vascular endothelial function and modulation of immune/inflammatory responses, which can antagonize the pathogenesis of hypertension through multiple pathways to lead a drop in BP theoretically. This theory has been preliminarily confirmed by several small sample-size studies. Therefore, this study intends to conduct a randomized controlled trial to further reveal the antihypertensive effect of LRIC and explore its potential mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-80 years；
2. Office blood pressure ≥130/80mmHg and<160/100mmHg; and 24-h ambulatory systolic/diastolic blood pressure ≥125/75mmHg;
3. Never taking antihypertensive drugs or have stopped taking antihypertensive drugs for more than one month;
4. Do not receive any antihypertensive drugs during the research;
5. Informed consent obtained from the subjects or their legally authorized representative.

Exclusion Criteria:

1. Secondary hypertension;
2. Patients who are taking antihypertensive drugs regularly;
3. Patients with contraindication for remote ischemic conditioning, such as vascular injury, soft tissue injury, orthopedic injury, or arm infection;
4. Patients with bleeding disorder;
5. Patients with atrial fibrillation or other severe arrhythmias；
6. Patients with prior myocardial infarction or stroke；
7. Patients with serious or unstable medical condition, such as severe liver or kidney dysfunction, heart failure, respiratory failure, malignant tumors, or autoimmune diseases;
8. Participation in another device or drug trial simultaneously;
9. Patients who are not suitable for this trial considered by researchers for other reasons.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Changes of average 24-h ambulatory systolic blood pressure. | From baseline to 4 weeks.
  Changes of average 24-h ambulatory systolic blood pressure from baseline to four weeks.

SECONDARY OUTCOMES:
Changes of average 24-h ambulatory diastolic blood pressure. | From baseline to 4 weeks.
  Changes of average 24-h ambulatory diastolic blood pressure from baseline to four weeks.
Changes of average daytime ambulatory systolic blood pressure. | From baseline to 4 weeks.
  Changes of average daytime ambulatory systolic blood pressure from baseline to four weeks.
Changes of average daytime ambulatory diastolic blood pressure. | From baseline to 4 weeks.
  Changes of average daytime ambulatory diastolic blood pressure from baseline to four weeks.
Changes of average night-time ambulatory systolic blood pressure. | From baseline to 4 weeks.
  Changes of average night-time ambulatory systolic blood pressure from baseline to four weeks.
Changes of average night-time ambulatory diastolic blood pressure. | From baseline to 4 weeks.
  Changes of average night-time ambulatory diastolic blood pressure from baseline to four weeks.
Changes of average 24-h heart rate. | From baseline to 4 weeks.
  Changes of average 24-h heart rate from baseline to four weeks.
Proportion of patients with average 24-h ambulatory systolic blood pressure reduction more than 5 mmHg. | From baseline to 4 weeks.
  Proportion of patients with average 24-h ambulatory systolic blood pressure reduction more than 5 mmHg.
Changes of office systolic blood pressure. | From baseline to 4 weeks.
  Changes of office systolic blood pressure from baseline to four weeks.
Changes of office diastolic blood pressure. | From baseline to 4 weeks.
  Changes of office diastolic blood pressure from baseline to four weeks.
Changes of vascular endothelium function(flow-mediated dilation , FMD) or arterial Stiffness(brachial-ankle pulse wave velocity, ba-PWV). | From baseline to 4 weeks.
  Changes of FMD or ba-PWV from baseline to four weeks.
Changes of blood biomarkers. | From baseline to 4 weeks.
  Changes of blood biomarkers which have been demonstrated to correlate with hypertension, such as NO、ET-1、IL-10、TNF-α、IL-1β、SDF-1α, from baseline to four weeks.
Adverse events related or not related to RIC treatment. | From baseline to 4 weeks.
  Adverse events related to RIC treatment, such as local edema, erythema, skin lesions of the arms, or adverse events not related to RIC treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, Principal Investigator — Xuanwu Hospital, Beijing
Locations (3):
- China (3):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Care Health Management Center, Beijing, Beijing Municipality
  - The 306 Hospital of People's Liberation Army, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao Y, Ren C, Li X, Yu W, Li S, Li H, Wang Y, Li D, Ren M, Ji X. Ischemic Conditioning Ameliorated Hypertension and Vascular Remodeling of Spontaneously Hypertensive Rat via Inflammatory Regulation. Aging Dis. 2021 Feb 1;12(1):116-131. doi: 10.14336/AD.2020.0320. eCollection 2021 Feb. PMID 33532132
- [Background] Tong XZ, Cui WF, Li Y, Su C, Shao YJ, Liang JW, Zhou ZT, Zhang CJ, Zhang JN, Zhang XY, Xia WH, Tao J. Chronic remote ischemic preconditioning-induced increase of circulating hSDF-1alpha level and its relation with reduction of blood pressure and protection endothelial function in hypertension. J Hum Hypertens. 2019 Dec;33(12):856-862. doi: 10.1038/s41371-018-0151-1. Epub 2019 Jan 10. PMID 30631131
- [Background] Madias JE. Sustained blood pressure lowering effect of twice daily remote ischemic conditioning sessions in a normotensive/prehypertensive subject. Int J Cardiol. 2015 Mar 1;182:392-4. doi: 10.1016/j.ijcard.2014.12.159. Epub 2015 Jan 3. No abstract available. PMID 25596469
- [Derived] Guo W, Zhao W, Li D, Jia H, Ren C, Li S, Zhao J, Yu B, Dong J, Guo R, Zhu K, Cao Y, Wang Y, Wang Y, Li Z, Wang Z, Wang D, Hou C, Hausenloy DJ, Chu X, Ji X. Chronic Remote Ischemic Conditioning on Mild Hypertension in the Absence of Antihypertensive Medication: A Multicenter, Randomized, Double-Blind, Proof-of-Concept Clinical Trial. Hypertension. 2023 Jun;80(6):1274-1282. doi: 10.1161/HYPERTENSIONAHA.122.20934. Epub 2023 Apr 10. PMID 37035920